CLINICAL TRIAL: NCT04553679
Title: Development of an Online Mindfulness Program for Stroke Survivors and Their Caregivers
Brief Title: Mindfulness After Stroke
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Carolee Winstein, Professor, University of Southern California
Other Study IDs: UP-20-00568
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Caregiver Burden
Keywords: Mindfulness; Rehabilitation; Caregiver; Attention to variability
MeSH Terms: conditions — Stroke; Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke survivors: Participants who have had a stroke
  Interventions: Behavioral: Mindfulness online intervention
- Caregivers: Participants who are caring for someone who have had a stroke
  Interventions: Behavioral: Mindfulness online intervention

INTERVENTIONS:
Behavioral: Mindfulness online intervention — A 3-week mindfulness intervention will be offered entirely online. The purpose of the intervention is: 1) to increase participants' mindfulness, and 2) to encourage participants to change their beliefs about the disability associated with stroke to improve their psychological state. Mindfulness refers to the act of being aware: aware of thoughts, aware of emotions, aware of physical sensations, aware of others. The intervention consists of educational texts, daily exercises, audio recordings and videos. Five different topics related to mindfulness will be introduced throughout the intervention.

SUMMARY:
The purpose of this study is to test the relevance, satisfaction and ease-of-use of an online mindfulness intervention among stroke survivors and their caregivers. Quality of life, depression, anxiety, stress and sleep quality will be assessed before, after and at 1 month after the intervention. After the intervention, participants' feedback about the usability and the satisfaction with the intervention and the online program will be gathered. Based on participants' feedback, changes to the intervention will be made to obtain a final version.

DETAILED DESCRIPTION:
The incidence of depression and anxiety is much higher in stroke survivors and their caregivers compared to age-matched peers. Previous work suggests that mindfulness delivered in an online format is promising for both individuals with neurological disorders and caregivers to improve quality of life and psychological well-being.

The overall objective of this project is to develop and refine an online mindfulness program that is perceived as relevant and user-friendly for stroke survivors and their caregivers. This project also aims to determine the potential impact of the mindfulness program on psychological well-being for stroke survivors and caregivers to guide the development of a future intervention study.

The process of development of the online mindfulness program will be iterative and will involve three phases: one development phase, one usability testing phase with end-users and one refinement phase.

Phase 1) The 3-week online mindfulness program will be adapted from the program developed for individuals with amyotrophic lateral sclerosis by mindfulness and stroke experts to ensure suitability and relevance for individuals with stroke.

Phase 2) A testing phase will be conducted remotely for both technical and clinical verification with 5-10 stroke survivors and 5-10 caregivers. Self-reported questionnaires about psychological well-being will be administered prior to and after the participation to the program and at a 1-month follow-up. After the program, a usability questionnaire and a semi-structured interview will be conducted to assess the usability of the mindfulness program and gather participants' feedback. For each group, differences prior to and after the mindfulness program will be assessed using a repeated measure analysis of variance. The transcribed verbatim of the semi-structured interview will be analyzed independently using thematic content analysis by 2 members of the research team.

Phase 3) Based on the results from Phase 2, modifications will be made to the online mindfulness program. If warranted, the testing phase will be replicated with a second cohort of participants.

This project will lead to the development of an online mindfulness program suitable for stroke survivors and their caregivers to improve quality of life and psychological well-being. This project will help guide the development of a planned intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke (for stroke survivors) or caregiver of someone who have had a stroke
* Ability to access Internet using a computer, a tablet and/or a smart phone
* Ability to provide informed consent
* Fluent in English

Exclusion Criteria:

* Severe language impairments
* Regular meditation or participation in a mindfulness program in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A convenience sample of 5-10 people with stroke and their caregivers will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolee Winstein, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Caregivers: Participants caring for someone who have had a stroke
Period: Overall Study
Arm/Group | Stroke Survivors | Caregivers
Started | 13 | 3
Completed | 11 | 2
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Caregiver only took part in the qualitative interview (no quantitative outcomes) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Caregivers: Participants who care for someone who have had a stroke
- Total: Total of all reporting groups
Arm/Group | Stroke Survivors | Caregivers | Total
Number analyzed (Participants) | 13 | 3 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant in the caregiver group did not receive the intervention, but participated to the qualitative interview to provide feedback about the program.
  years | 65.1 (12.1) | 59.7 (21.5) | 64.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 9 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 1 | 9
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Stroke Impact Scale
Description: Quality of life and impact of stroke after the intervention. The Stroke Impact Scale is a 59-item measure and is divided in 8 domains. Scores range from 0-100 (with higher score showing better quality of life and lower stroke impact).
Time Frame: from baseline to 3 weeks
Population: The Stroke Impact Scale is a measure of stroke severity. It was not administered to caregivers. Two stroke survivors did not complete the post-intervention measurement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stroke Survivors
Number analyzed (Participants) | 11
score on a scale | 2.3 (24.3)

2. Secondary Outcome: Change in Hospital Anxiety and Depression Scale
Description: The Hospital Anxiety and Depression Scale (HADS) is a 14-item scale with 7 items each for anxiety and depression subscales. Each item is scored from 0 to 3, with higher scores indicating higher anxiety or depressive symptoms. Anxiety and depression with scores ranging from 0 (no depression/anxiety) to 21 (severe depressive/anxious symptoms).
Time Frame: from baseline to 3 weeks
Population: Two stroke survivors did not complete the post-intervention measurement. One caregiver group did not receive the intervention (only did the qualitative portion of the study).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stroke Survivors | Caregivers
Number analyzed (Participants) | 11 | 2
score on a scale | 0.9 (3.5) | 5 (1.4)

3. Secondary Outcome: Change in National Institute of Health Perceived Stress Survey
Description: 10-item self-reported measure assessing perceived stress. Scores range from 10 to 50, with higher scores indicating greater levels of perceived stress.
Time Frame: from baseline to 3 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Caregivers: Participants who care for a stroke survivors
Arm/Group | Stroke Survivors | Caregivers
Number analyzed (Participants) | 11 | 2
score on a scale | 1.1 (5.1) | 4.5 (3.5)

4. Secondary Outcome: Change in Single-Item Sleep Quality Scale
Description: 1-item sleep quality scale ranging from 1 to 10. Higher scores indicate better sleep quality.
Time Frame: from baseline to 3 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stroke Survivors | Caregivers
Number analyzed (Participants) | 11 | 2
units on a scale | 0.9 (2.1) | 4 (1.4)

5. Secondary Outcome: Change in World Health Organization Quality of Life-bref
Description: The World Health Organization Quality of Life-BREF (WHOQOL-BREF) comprises 26 questions from 4 domains about health and well-being: 1) Physical health (e.g., Activities of daily living, Mobility, Fatigue, etc.), 2) Psychological (e.g., Negative/positive feelings, Self-esteem, Spirituality, etc.), 3) Social relationships (e.g., Personal relationships, Social support, Sexual activity), 4) Environment (e.g., financial resources, home environment, opportunities for leisures, etc.). The scores are transformed on a scale from 0-100. Higher scores indicate better perceived health and well-being.
  Outcome measure only administered to caregivers.
Time Frame: from baseline to 3 weeks
Population: One caregiver group did not receive the intervention (only did the qualitative portion of the study).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 2
score on a scale | 6.25 (4.7)

6. Secondary Outcome: Adapted Post-Study System Usability Questionnaire
Description: The adapted Post-Study System Usability Questionnaire (PSSUQ) consists of 5 questions on perceived satisfaction with the online platform used to host the program. Each question is scored on a 7-point Likert scale from 1 (Strongly Agree) to 7 (Strongly Disagree) for a total score of 35. Higher scores indicate lower usability.
Time Frame: 3 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stroke Survivors | Caregivers
Number analyzed (Participants) | 11 | 2
score on a scale | 14.3 (7.9) | 24.5 (12.0)

7. Secondary Outcome: Change in Zarit Burden Interview
Description: The Zarit Burden Interview includes 22 questions about caregiver burden rated from 0 (never) to 4 (nearly always). Scores range from 0-88 with higher scores indicating greater burden.
  Measure administered only to participants in the caregiver group.
Time Frame: from baseline to 3 weeks
Population: One caregiver group did not receive the intervention (only did the qualitative portion of the study).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 2
score on a scale | 3 (9.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study period (up to 1 month post-intervention).
Description: The clinicaltrials.gov definition was used.
Arm/Group | Stroke Survivors | Caregivers
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/3
Other Adverse Events (participants affected / at risk) | 0/13 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stroke Survivors (N=13) | Caregivers (N=3)
Moderate Adverse Event (Shoulder pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Polymyalgia rheumatica diagnosed during the participation to the study

LIMITATIONS AND CAVEATS:
Our sample was small and heterogenous. This study was not powered to detect changes in the self-reported measures, but it provided guidance on the selection of outcome measures for a larger intervention study. The possibility of a social desirability bias is not excluded since participants may have wanted to please the researchers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT04553679/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT04553679/SAP_001.pdf